CLINICAL TRIAL: NCT03615118
Title: AniMovil mHealth Support for Depression Management in a Low-Income Country
Acronym: AniMovil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Universidad de Los Andes, Bogota, Colombia (Unknown)
Responsible Party: Principal Investigator, John Piette, VA Senior Research Career Scientist and Professor of Health Behavior Health Education, Public Health, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 15-PAF05075
Record Dates: First submitted 2018-07-13; First posted 2018-08-03 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients randomized to the intervention group will receive the AniMóvil intervention, including: the Sentirse Mejor manual that patients can refer to for information about CBT and skill practice, weekly IVR depression symptom assessments and psychoeducational messages, daily SMS mood monitoring and CBT reinforcement messages, and CHW telephone CBT sessions in the event of elevated PHQ-9 scores during the study. CHWs will use information from patients' IVR/SMS monitoring to support intervention-group patients' depression self-management under close supervision from their mental health specialist supervisor. Intervention patients will be part of a 'stepped' intervention based on the severity of their depression upon entry into the program and assessment throughout the intervention.
  Interventions: Other: IVR/SMS
- Enhanced Usual Care (Active Comparator): Enhanced usual care patients will receive usual care, including the Sentirse Mejor manual developed by the research team in conjunction with local Ministries of Mental Health and tailored by the study team, emphasizing CBT principles, and daily SMS messages asking participants to report their mood on a 1 to 9 scale. Enhanced usual care group patients who report mood scores of 1 or 2 (worst scores) for at least 3 days per week and 3 consecutive weeks will be called by the Community health worker and referred to the national program office for depression services support - a free service available to all citizens diagnosed with depression. Enhanced usual care patients will be part of a 'stepped' program based on the severity of their depression upon entry into the program and assessment throughout the intervention.
  Interventions: Other: SMS

INTERVENTIONS:
Other: IVR/SMS — Daily SMS messages asking participants to report their mood on a 1 to 9 scale; An automated phone system for monitoring and improving self-care and health outcomes
  Arms: Intervention
Other: SMS — Daily SMS messages asking participants to report their mood on a 1 to 9 scale
  Arms: Enhanced Usual Care

SUMMARY:
Depression is a huge public health problem in low and middle-income countries (LMICs). Mental health care systems in most LMICs are extremely limited, impeding the dissemination of WHO-recommended models for improving care via "task-shifting" services to community health workers (CHWs) who deliver evidence-based treatments such as cognitive behavioral therapy (CBT). This comprehensive intervention will use IVR and text messaging (SMS) to support effective depression care. Intervention patients will receive weekly automated (IVR) calls and daily text messages (SMS) throughout the 12 week intervention. Patients with more severe depression will receive up to 12 weekly CHW-delivered telephone CBT sessions, based on WHO recommendations and a treatment model developed and tested in India. CHWs will use patients' IVR contacts to enhance psychoeducation and they will use SMS plus web-based reports based on patients' IVR calls to identify individuals needing additional follow-up. The CHWs' clinical supervisor will use SMS messages to CHWs to reinforce best practices and monitor service delivery.

Patients will be enrolled from Colombian clinics associated with the Universidad de Los Andes in Bogota, Colombia. 114 patients will be randomized to either a usual enhanced care or intervention group. Intervention group patients will receive weekly automated (IVR) calls and daily text messages throughout the duration of the 12 week intervention. Patients with more severe depression will receive up to 12 weekly CHW-delivered telephone CBT sessions, based on WHO recommendations and a treatment model developed and tested in India. CHWs will use patients' IVR contacts to enhance psychoeducation and they will use SMS plus web-based reports based on patients' IVR calls to identify individuals needing additional follow-up. The CHWs' clinical supervisor will use SMS messages to CHWs to reinforce best practices and monitor service delivery. Program components will be modified to fit the local culture and clinical environment via iterative engagement of health professionals and patients with depression.

Those patients in usual enhanced care will receive the study manual and daily text messages and feedback throughout the duration of the program. Patients in the enhanced usual care group who present with more severe depression will be referred to the national program office for depression services support - a free service available to all citizens diagnosed with depression.

ELIGIBILITY:
Inclusion Criteria:

* A score of 10+ on the Spanish-validated version of the PHQ-9

Exclusion Criteria:

* Less than a 6-month life expectancy
* A history of psychiatric hospitalization or bipolar disorder
* A substance use disorder or cognitive impairment

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Severity of depression symptoms, as measured by Patient Health Questionnaire, 9 item (PHQ9) | Change in PHQ scores at Baseline and 3 month follow-up
  Depressive symptom severity. Min score=0, Max score=27. 0=not depressed, 27=severe depression.

SECONDARY OUTCOMES:
Health related quality of life as measured by Short Form Survey (SF12) | Change in SF12 score at Baseline and 3 month follow-up
  The SF-12 is composed of 12 questions, selected from the SF-36 Health Survey (Ware, Kosinski, and Keller, 1996). The 12 questions are combined, scored, and weighted, assessing mental and physical functioning and overall health-related-quality of life.
Sheehan Disability Scale (SDS) | Change in score at Baseline and 3 month follow-up
  The SDS is a brief, 5-item self-report tool that assesses functional impairment in work/school, social life, and family life. 0=not at all, 1-3=mild, 4-6=moderate, 7-9=marked, 10=extremely. Total score 0-30 (0 unimpaired, 30 highly impaired). Questions are broken into 3 assessed categories: Work/school (0-10); Social life (0-10); Family life/home responsibilities (0-10). Scoring: Scores of ≥5 on any of the 3 scales indicate a high score, and high scores are associated with significant functional impairment.
Daily mood ratings | Changes in Daily mood scores between days 1-90
  Daily mood rating on a 1-9 scale reported via SMS. Daily mood score of 1 indicates a low mood, where as 9 indicates a high or positive mood.

CONTACTS AND LOCATIONS:
Overall Officials: John Piette, PhD, Principal Investigator — University of Michigan
Locations (1):
- Hospital San Jose, Bogotá, Colombia